CLINICAL TRIAL: NCT02735382
Title: Transforming the Treatment of Tobacco Use in Health Care: Seizing the Potential of the Electronic Health Record to Deliver Comprehensive Chronic Care Treatment for Smoking: Study 1: the EHR and Fax Referral Study
Brief Title: EHR-Based and Fax-Based Referral to a Tobacco Quitline: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0844; 1R35CA197573-01 (NIH)
Record Dates: First submitted 2016-04-01; First posted 2016-04-12 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Tobacco Use Cessation; Tobacco Smoking
Keywords: Translational Medical Research; Clinical Practice Guidelines; Electronic Health Records; Smoking; Tobacco; Quitline
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Smoking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EHR-based referral to quit line (Experimental): Clinics will use an EHR-based fully-electronic HIPAA-compliant tool to refer their adult patients who use tobacco to the telephone tobacco quitline for tobacco cessation counseling and medication.
  Intervention: Behavioral: Tobacco quitline EHR referral
  Interventions: Behavioral: Tobacco quitline EHR referral
- Fax-based referral to quit line (Active Comparator): Clinics will use a paper fax tool to refer their adult patients who use tobacco to the telephone tobacco quitline for tobacco cessation counseling and medication.
  Intervention: Behavioral: Tobacco quitline Fax referral
  Interventions: Behavioral: Tobacco quitline Fax referral
- EHR-based Clinic Staff (Experimental): Clinics will use an EHR-based fully-electronic HIPAA-compliant tool to refer their adult patients who use tobacco to the telephone tobacco quitline for tobacco cessation counseling and medication. Staff in these clinics will complete surveys to address Aim 4 of the study.
  Interventions: Behavioral: Tobacco quitline EHR referral
- Fax-based referral to quit line Clinic Staff (Active Comparator): Clinics will use a paper fax tool to refer their adult patients who use tobacco to the telephone tobacco quitline for tobacco cessation counseling and medication. Staff in these clinics will complete surveys to address Aim 4 of the study.
  Interventions: Behavioral: Tobacco quitline Fax referral

INTERVENTIONS:
Behavioral: Tobacco quitline EHR referral — Using an EHR-based referral to the tobacco quitline from primary care outpatient clinics.
  Arms: EHR-based Clinic Staff; EHR-based referral to quit line
Behavioral: Tobacco quitline Fax referral — Using an Fax--based referral to the tobacco quitline from primary care outpatient clinics.
  Arms: Fax-based referral to quit line; Fax-based referral to quit line Clinic Staff

SUMMARY:
This study is designed to assess whether completely electronic, HIPAA-compliant, EHR-based, closed-loop referrals for tobacco cessation from primary care clinics to a state telephone tobacco quitline service can increase the number/percentage of adult tobacco users receiving evidence-based tobacco dependence treatment when compared to paper-based fax referrals. This study also will survey clinic staff to evaluate satisfaction with the referral process.

DETAILED DESCRIPTION:
Aim 1: To evaluate the rates of referral of tobacco users visiting primary care clinics to the WTQL, comparing those who were referred via an EHR-based electronic referral system vs. those referred via a manual paper fax referral system. Analyses will address the change in rates of referrals from pre- to post-intervention and the trajectory of referral post-intervention and will reflect per clinic rates.

Aim 2: To evaluate the rates of quality referrals of tobacco users visiting primary care clinics to the WTQL, comparing those who were referred via an EHR-based electronic referral system vs. those referred via a manual paper fax referral system (quality referrals are defined as ones that result in individuals who enroll in and receive WTQL counseling and/or medication treatment services). Analyses will address the change in referrals from pre- to post-intervention and will reflect per clinic rates.

Aim 3: To examine variation in referral rates across clinics to test the hypothesis that the eReferral system will result in greater consistency in referral in addition to higher rates of referral. Qualitative methods will be used to understand the sources of variation.

Aim 4: To assess clinician and staff satisfaction with the eReferral and paper fax referral systems via self-report questionnaires.

Aim 5: To evaluate smoking abstinence rates of tobacco users who were referred to and accepted services from the WTQL, comparing those who were referred via an EHR-based referral system vs. those referred via a manual paper fax referral system.

ELIGIBILITY:
Clinic Eligibility:

Inclusion Criteria:

* The presence of discrete primary care clinical services within the clinic (defined as general internal medicine or family medicine clinical services);
* At least three primary care clinician providers in the clinic (physicians or nurse practitioners/physician assistants who see patients independently of a physician);
* A total primary care clinical volume of at least 60 patients each week;
* An existing EHR requirement for staff to document tobacco use status including smoking status on all adult patients visiting the clinic at every visit;
* A capacity to enumerate patient visit information including adult patients/month and adult tobacco users/month by clinician and by clinic;
* A willingness to participate in the proposed research;
* A lead physician or a clinic manager on site who agree to serve as a clinic champion for the project;
* Prior use of the fax referral system to refer patients to the Wisconsin Tobacco Quit Line with use data available for the 12 months prior to study launch;
* A willingness to accept random assignment to either of the two experimental conditions.

Exclusion Criteria:

* Those clinics not meeting the above criteria (e.g. too small, limited EHR capacity).

(Note: In this study, the clinics are the "subjects" under study. The patients that will be referred by the clinic to the Wisconsin Tobacco Quit Line will be least 18 years old and Cigarette smokers)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14930 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fiore, MD, MPH, MBA, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zehner ME, Kirsch JA, Adsit RT, Gorrilla A, Hayden K, Skora A, Rosenblum M, Baker TB, Fiore MC, McCarthy DE. Electronic health record closed-loop referral ("eReferral") to a state tobacco quitline: a retrospective case study of primary care implementation challenges and adaptations. Implement Sci Commun. 2022 Oct 8;3(1):107. doi: 10.1186/s43058-022-00357-4. PMID 36209149
- [Derived] Fiore M, Adsit R, Zehner M, McCarthy D, Lundsten S, Hartlaub P, Mahr T, Gorrilla A, Skora A, Baker T. An electronic health record-based interoperable eReferral system to enhance smoking Quitline treatment in primary care. J Am Med Inform Assoc. 2019 Aug 1;26(8-9):778-786. doi: 10.1093/jamia/ocz044. PMID 31089727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This cluster randomized clinical trial was conducted in 23 primary care clinics, representing 2 health systems in Wisconsin, randomized to eReferral (intervention; n = 11) or Fax-to-Quit (usual care; n = 12). All participants were adult patients attending visits at their primary care clinics.
Groups:
- EHR-based Referral to Quit Line: Clinics will use an EHR-based fully-electronic HIPAA-compliant tool to refer their adult patients who use tobacco to the telephone tobacco quitline for tobacco cessation counseling and medication.
  Intervention: Behavioral: Tobacco quitline EHR referral
  Tobacco quitline EHR referral: Using an EHR-based referral to the tobacco quitline from primary care outpatient clinics.
- Fax-based Referral to Quit Line: Clinics will use a paper fax tool to refer their adult patients who use tobacco to the telephone tobacco quitline for tobacco cessation counseling and medication.
  Intervention: Behavioral: Tobacco quitline Fax referral
  Tobacco quitline Fax referral: Using an Fax--based referral to the tobacco quitline from primary care outpatient clinics.
- EHR-based Referral to Quit Line Clinic Staff: Staff in these clinics that use EHR-based referral to the quit line will complete surveys to address Aim 4 of the study.
- Fax-based Referral to Quit Line Clinic Staff: Staff in these clinics that use Fax-based referral to the quit line will complete surveys to address Aim 4 of the study.
Period: Overall Study
Arm/Group | EHR-based Referral to Quit Line | Fax-based Referral to Quit Line | EHR-based Referral to Quit Line Clinic Staff | Fax-based Referral to Quit Line Clinic Staff
Started | 7481 | 7155 | 184 | 110
Completed | 7481 | 7155 | 184 | 110
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EHR-based Referral to Quit Line | Fax-based Referral to Quit Line | EHR-based Clinic Staff | Fax-based Referral to Quit Line Clinic Staff | Total
Number analyzed (Participants) | 7481 | 7155 | 184 | 110 | 14930
Age, Continuous [Mean (Full Range); unit: years] — Population: Clinic surveys were anonymous and, as such, no demographic information was collected.
  years
    number analyzed (Participants) | 7481 | 7155 | 0 | 0 | 14636
    (all) | 50.0 [18 to 90] | 48.8 [18 to 90] |  |  | 49.4 [18 to 90]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 0 | 0 | 0 | 0 | 0
  Unknown | 7481 | 7155 | 184 | 110 | 14930
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5712 | 5682 | 0 | 0 | 11394
  African American | 1631 | 1142 | 0 | 0 | 2773
  Other | 78 | 106 | 0 | 0 | 184
  Unknown | 60 | 225 | 184 | 110 | 579
Region of Enrollment [Number; unit: participants]
  United States | 7481 | 7155 | 184 | 110 | 14930

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Referred
Description: EHR-based vs. Fax-based rates of referral of adult tobacco users visiting primary care clinics to the tobacco quitline. The rate of referral will be determined by the ratio of total referrals to total smokers identified in the clinic's EHR over a period of 6 months of study observation.
Time Frame: Rates come from cumulative data collected over the course of 6 months.
Population: Participant data were derived from EHR records.
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Referral to Quit Line | Fax-based Referral to Quit Line
Number analyzed (Participants) | 7481 | 7155
Participants | 1380 | 331
Statistical Analysis 1: Comparison: EHR-based Referral to Quit Line vs Fax-based Referral to Quit Line; Test type: Superiority; p < .0001, Chi-squared, Corrected; Odds Ratio (OR) = 4.663, 95% CI 2-sided [4.116 to 5.283]

2. Secondary Outcome: Number of Participants Meeting Criteria for Quality Referral
Description: To evaluate the rates of quality referrals of tobacco users visiting primary care clinics to the tobacco quitline. Quality referrals are defined as ones that result in individuals who enroll in and receive tobacco quit line services.
Time Frame: Rates come from cumulative data collected over the course of 6 months.
Population: Participant data were derived from Quit Line records.
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Referral to Quit Line | Fax-based Referral to Quit Line
Number analyzed (Participants) | 7481 | 7155
Participants | 400 | 121
Statistical Analysis 1: Comparison: EHR-based Referral to Quit Line vs Fax-based Referral to Quit Line; Test type: Superiority; p < .0001, Chi-squared, Corrected; Odds Ratio (OR) = 3.284, 95% CI 2-sided [2.672 to 4.035]

3. Secondary Outcome: Number of Participants Self-reporting Smoking Abstinence
Description: To evaluate smoking abstinence rates of tobacco users who were referred to and accepted services from the WTQL, comparing those who were referred via an EHR-based referral system vs. those referred via a manual paper fax referral system.
Time Frame: 7-day point prevalence smoking outcomes at 4-months after participant registration with the WI Tobacco Quit Line.
Population: Participant data were derived from Quit Line records.
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Referral to Quit Line | Fax-based Referral to Quit Line
Number analyzed (Participants) | 7481 | 7155
Participants | 34 | 14
Statistical Analysis 1: Comparison: EHR-based Referral to Quit Line vs Fax-based Referral to Quit Line; Test type: Superiority; p = .8438, Chi-squared, Corrected; Odds Ratio (OR) = 0.885, 95% CI 2-sided [0.420 to 1.698]

4. Secondary Outcome: Change in Global Staff Satisfaction With the Referral Intervention
Description: In order to assess clinician and staff satisfaction with the eReferral and paper-based referral systems, a single-item "The steps I need to take to address my patients' tobacco use are efficient and well designed" was administered to healthcare system clinical staff. The response format was 1 = Strongly disagree; 2 = Disagree; 3 = Mildly disagree; 4 = Feel neutral; 5 = Mildly agree; 6 = Agree; 7 = Strongly agree. Higher scores indicate greater satisfaction with the assigned intervention (EHR-based vs Fax-based referral systems). The item is not part of any existing validated scale and was created for purposes of the project; this item was selected from a larger set of items and determined to be the most appropriate measure of overall staff satisfaction.
Time Frame: Satisfaction measures will be surveyed at baseline and at 6 months and reported as a single change score
Population: Clinic staff in the study clinics.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EHR-based Referral to Quit Line Clinic Staff | Fax-based Referral to Quit Line Clinic Staff
Number analyzed (Participants) | 184 | 110
units on a scale | 0.76 (1.37) | 0.32 (1.28)
Statistical Analysis 1: Comparison: EHR-based Referral to Quit Line Clinic Staff vs Fax-based Referral to Quit Line Clinic Staff; A change score from baseline to 6-months was computed and served as the data to be analyzed in the t-test of group differences; Test type: Superiority; p = .007, t-test, 2 sided; df=292; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [0.123 to 0.757], Standard Error of Mean 0.161

ADVERSE EVENTS:
Time Frame: Adverse event data not collected. This was an EHR-based study.
Description: Adverse event data not collected. This was an EHR-based study.
Arm/Group | EHR-based Referral to Quit Line | Fax-based Referral to Quit Line | EHR-based Referral to Quit Line Clinic Staff | Fax-based Referral to Quit Line Clinic Staff
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT02735382/Prot_SAP_000.pdf